CLINICAL TRIAL: NCT07195032
Title: Safety and Efficacy of Measles, Mumps, Rubella Vaccination in Pediatric Heart Transplantation Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Victoria Blazek, Clinical Pharmacy Specialist, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003689
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Heart Transplant Infection Prevention
Keywords: Measles; Mumps; Rubella; Live vaccine; Heart transplant
MeSH Terms: conditions — Measles; Mumps; Rubella | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Measles, Mumps, Rubella Vaccination (Experimental): Patients receiving MMR vaccination due to no historical vaccine OR a seronegativity for measles
  Interventions: Drug: Commercial measles, mumps, and rubella (MMR) vaccine

INTERVENTIONS:
Drug: Commercial measles, mumps, and rubella (MMR) vaccine — Participants will receive the commercial MMR vaccine if they are deemed eligible for the study.

SUMMARY:
The study is an interventional, non-randomized assessment of safety and efficacy of live Measles, Mumps and Rubella (MMR) vaccine in subjects aged 12-months to 17 years who have undergone heart transplantation. Subjects who provide permission/assent will receive the commercial MMR vaccine according to product indication and labeling.

ELIGIBILITY:
Inclusion Criteria:

* Received a heart transplant
* At least 1 year after transplant
* At least 1 year after antibody-mediated rejection treatment (intravenous immune globulin, rituximab, bortezomib, plasmapheresis, carfilzomib, eculizumab, daratumumab)
* At least 1 year from anti-thymocyte globulin
* At least 6 months after pulse dose steroid treatment or basiliximab treatment
* No history of MMR vaccination OR History of MMR vaccination but seronegativity for measles at time of inclusion
* Clinically well

Exclusion Criteria:

* History of repeated infections necessitating adjustment in immunosuppression to non-standard regimen, including single agent immunosuppression and modified trough levels.
* History of anaphylactic reaction to MMR vaccination

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2027-09-11 (Estimated); Study Completion 2027-09-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experience adverse reactions to the measles, mumps, and rubella vaccination | Between 0-240 days after vaccine administration
  Patients will be screened for adverse reactions following vaccine administration
Number of participants with resultant initial seropositivity against measles after vaccination | Between 60-240 days after vaccine administration.
  Serologic response will be measured after vaccine administration.

SECONDARY OUTCOMES:
Number of participants who experience prolonged seropositivity after vaccine administration | Minimum of 365 days after vaccine administration
  Serologic response will be tested at least 365 days after final vaccine administration

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Blazek, PharmD, BCPPS, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided